CLINICAL TRIAL: NCT02841800
Title: Intra-luminal Radiofrequency Ablation for Inoperable Malignant Biliary Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201604030DIPD
Record Dates: First submitted 2016-07-19; First posted 2016-07-22 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Liver Cancer; Bile Duct Cancer; Pancreatic Cancer
Keywords: radiofrequency ablation; malignant biliary stenosis
MeSH Terms: conditions — Liver Neoplasms; Bile Duct Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intra-luminal radiofrequency ablation (Experimental): Intra-luminal radiofrequency ablation Admission for endoscopic retrograde cholangiopancreatography (ERCP) and stent placement after radiofrequency ablation. ERCP should be performed for 2 times with an interval of two months.
  Interventions: Device: 'Intra-luminal radiofrequency ablation (Habib EndoHPB)

INTERVENTIONS:
Device: 'Intra-luminal radiofrequency ablation (Habib EndoHPB) — endobiliary radiofrequency ablation device

SUMMARY:
Only a small proportion of patients with biliary obstruction caused by hepatopancreatobiliary malignancies are suitable for surgical resection. Therefore, most patients with malignant biliary obstruction will need palliation of their obstructive jaundice to relieve the symptoms and prevent life threatening complications such as biliary sepsis. The endoscopic or percutaneous/transhepatic routes, such as endoscopic retrograde cholangiopancreatography (ERCP) and percutaneous transhepatic cholangiography (PTC), and stents are accepted approaches for the relief of jaundice in malignant biliary obstruction. Improvement in the bilirubin level is also essential before palliative chemotherapy is considered in these patients. However, tumor ingrowth still remains a major cause of obstruction. In this trial, the investigators will use HabibTM EndoHPB (EMcision Ltd., UK) catheter which was used for the endobiliary radiofrequency ablation (RFA) treatment as a form of neoadjuvant therapy in hepatopancreatobiliary adenocarcinoma.

DETAILED DESCRIPTION:
The HabibTM EndoHPB (EMcision Ltd., UK) catheter which was used for the endobiliary radiofrequency ablation (RFA) treatment is an endoscopic bipolar catheter designed to ablate tissue in malignant tumors within luminal structures. HabibTM EndoHPB has Food and Drug Administration (FDA) and European Conformity approval for such indications. It has also approved by Ministry of Health and Welfare in 2016. In this study, the investigators will perform intra-luminal RFA for 20 inoperable patients with malignant biliary stenosis. HabibTM EndoHPB will be deployed via an endoscopic retrograde cholangiopancreatography (ERCP) route. By using radiofrequency energy to heat the tissue in the duct prior to insertion of the stent, the surrounding tissue becomes coagulated and this may delay tumor growth and the time before the stent lumen becomes occluded. If stent occlusion occurs in a participant during the follow up period, the participant will be reassessed and investigations will be used to determine cause of stent occlusion and whether it is appropriate to repeat RFA treatment. The aim will be to detect an improvement in survival and safety in the treated patients compared to patient receiving palliative treatment recorded in literatures.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible for this study:

  1. 20 Years and older.
  2. The diagnosis of hepatopancreaticobiliary cancers with pathologic proven, and the diagnosis of hepatopancreaticobiliary cancers will be made by pathology / cytology or according to the American Association for the Study of Liver Diseases (AASLD) (2010) diagnostic criteria.
  3. Participant unsuitable for surgical resection. Criteria for unresectability being based on metastatic disease or locally advanced.
  4. Eastern Cooperative Oncology Group (ECOG) score of 0-1.
  5. American Society of Anaesthesiologists (ASA) score ≤ 3.
  6. Karnofsky score >30.
  7. Jaundice (bilirubin level over 10 mg/dL). Alanine transaminase (ALT) and aspartate transaminase (AST) < 5 x upper limit of normal.
  8. Prothrombin time (PT)- international normalized ratio (INR) ≦ 2.0. Platelet count ≥ 100 K/Μl.
  9. Expected to survive more than 3 months.

Exclusion Criteria:

* Patients presenting with any of the following will not be enrolled into this study:

  1. Under the age of 20 years old.
  2. Women who are pregnant or women of child-bearing potential who are not using an acceptable method of contraception.
  3. Known history of human immunodeficiency virus (HIV) infection.
  4. Patients who have any serious or systemic disease that is not a good fit for this test.
  5. Tumor occupying more than 50% of liver parenchyma
  6. Any active metal implanted device (eg Pacemaker).
  7. Guidewire cannot pass through the bile duct stenosis.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-06; Primary Completion 2018-08-30 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
survival benefit | up to 3 months
  whether survival benefit is conferred to patients in the study at 3 months
survival benefit | up to 6 months
  whether survival benefit is conferred to patients in the study at 6 months
survival benefit | up to 12 months
  whether survival benefit is conferred to patients in the study at 12 months

SECONDARY OUTCOMES:
the recurrence of bile duct obstruction and jaundice | up to 3 years
  To analyze the recurrence of bile duct obstruction and jaundice.
potential treatment-related complications | up to 3 years
  To analyze potential treatment-related complications
repeated biliary interventions | up to 3 years
  To analyze the number of repeated biliary interventions

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, MD, PhD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No